CLINICAL TRIAL: NCT02602730
Title: Internet-Based Nonsmoking Program for Postpartum Women
Acronym: PostPartum_2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Principal Investigator, Susan Schroeder, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SBIR80RR-II; R44CA112739-01A2 (NIH)
Record Dates: First submitted 2015-01-02; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Cigarette Smoking; Smoking, Tobacco
Keywords: Cigarette smoking; Smoking, Tobacco; postpartum; internet; interactive; coach
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Break the Chain (Experimental): Access during the evaluation study period to an Internet smoking cessation intervention that included digital coaching messages sent at prescribed times during the participant's quit process and as needed in response to participant questions or comments.
  Interventions: Behavioral: Break the Chain
- Clearing the Air PDF (Active Comparator): Control users were e-mailed a copy of the National Cancer Institute's PDF smoking cessation booklet, "Clearing the Air."
  Interventions: Behavioral: Clearing the Air

INTERVENTIONS:
Behavioral: Break the Chain — Internet-based smoking cessation intervention designed for general population smokers with targeted materials for pregnant women. The program included a digital coaching component delivered via email at specific points as the user progresses through his/her quit process. Program content is based on Department of Health and Human Services Clinical Practice Guidelines for Treating Tobacco Use and Dependence.
  Arms: Break the Chain
Behavioral: Clearing the Air — PDF version of smoking cessation booklet from National Cancer Institute.
  Arms: Clearing the Air PDF

SUMMARY:
This project developed and evaluated an Internet-based interactive program with digital coaching designed to assist two groups of smokers in quitting smoking: (1) pregnant smokers and (2) general-population smokers (i.e., men and non-pregnant women). Program content was based on the U.S. Department of Health and Human Services Clinical Practice Guidelines, "Treating Tobacco Use and Dependence: 2008 Update" (Fiore et al., 2008) and input from project consultants.

DETAILED DESCRIPTION:
The "Break the Chain" program is an online smoking cessation intervention that incorporated strategic message construction based on behavior change constructs, interactive exercises, and digitial coaching support to engage the user in their smoking behavior change. The Expanded Theory of Reasoned Action (ETRA) (Fishbein, 1999, 2000) provides the theoretical foundation for the content. Intervention components include: (1) interactive check-ins, (2) content modules and interactive smoking cessation tools, (3) digital coaching, and (4) online social media (i.e., article feed).

Content modules included: Benefits of quitting, Making a plan for quitting, Boosting your support system, Planning for cravings and tempting situations, Managing stress and mood, Managing your weight, and Becoming an ex-smoker. Tailored information within each module was presented to the user based on responses to initial assessment questions and interactive check-ins (e.g., readiness to quit, pregnancy status, previous quit attempts, self-efficacy for quitting, worry about weight gain). Interactive tools presented within the logical flow of the modules included a Reasons for Quitting questionnaire, Pros and Cons of Quitting tool (decisional balance), Nicotine Dependence quiz, a Pharmacological Aid Decision tool, and a Quit Meter. Content was entirely text-based.

Within-program coach-generated and program-generated messages provided cessation tips and information. Digital coaching contacts were timed and tailored to the user's smoking status, health history, pregnancy status (if appropriate), and timing of quit day. The coaching messages prompted the user to engage more fully with the website by presenting hyperlinks to pertinent smoking cessation information or strategies in the program. A computer algorithm controlled the timing of the messages to each user. Users were invited to contact their coach via in-program message at any time with questions or concerns about smoking cessation strategies. A coaching interface allowed a health coach to view user information as the user progressed through the program and developed his/her quit plan. The coaching interface was also the platform through which the coach managed communication with each user.

ELIGIBILITY:
Inclusion criteria for pregnant:

* 18 years or older
* Between 8 and 32 weeks pregnant
* Currently smoking, trying to quit, or quit smoking within last 2 months
* Able to speak and read English
* Have access to high-speed or DSL Internet and email for the duration of the study.

Inclusion criteria for general population participants:

* Male or female not pregnant
* 18 years or older
* Currently smoking, trying to quit, or quit smoking within last 2 months
* Able to speak and read English
* Have access to high-speed or DSL Internet and email for the duration of the study

Exclusion critieria:

* Men and women under age 18 were excluded.
* Women who were pregnant but whose pregnancy did not fit within the specified time frame were excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of cigarettes smoked in the last 7 days | 10 months
  Smoking cessation as measured by number of cigarettes smoked in the last 7 days. We will use an intent-to-treat statistical analysis, a conservative approach that classifies all non-responders as smokers.

SECONDARY OUTCOMES:
Change from baseline in knowledge of impact of smoking cessation | 10 months
  Pregnant smokers only: Eight knowledge items assess post-natal impact (e.g., Smoking during pregnancy increases chances of having a child who develops asthma); seven items assess infant impact (e.g., Exposing an infant to smoke in the home increases the chances the baby will wake up at night more than usual); eight items assessed infant health risk (e.g., Babies exposed to secondhand smoke have increased chances of having learning disabilities). Response options were a "true" and "false" format scored to reflect the proportion of items answered correct in each domain. The seriousness of infant health issues related to smoking was assessed with five items (e.g., A baby born with lower than normal weight - low birth weight baby) with a five-point response option (1=not at all serious, 5=extremely serious). A mean score was computed and it showed good reliability (alpha = .82).
Change from baseline in self-efficacy to quit smoking | 10 months
  Six self-efficacy items (e.g., How confident are you that you could quit and stay quit) were assessed of all smokers. Each item had a five-point response option (1=not at all confident, 5=extremely confident) and showed good reliability (alpha=.86).
Change from baseline in attitudes about smoking cessation | 10 months
  Five attitude items (e.g., Knowing the right way to ask for help from family and friends when I'm quitting is important) were assessed of all smokers. Each item had a five-point response option (1=not at all important, 5=extremely important) and showed adequate reliability (alpha=.77).
Change from baseline in behavioral intentions about smoking cessation | 10 months
  Five intention items (e.g., How likely is it that you will avoid every situation where you will be tempted to smoke) were assessed of all smokers. Each item had a five-point response option (1=not at all likely, 5=extremely likely) and showed adequate reliability (alpha = .79).
Program satisfaction | 4-week posttest
  Seven program satisfaction items were assessed of as rated by the treatment participants at the T2 assessment. Treatment participants were also asked how likely they would be to recommend the program to a friend and/or family member.
User rating of system usability | 4-week posttest
  All treatment participants were asked how much they agreed or disagreed with program usability statements (see Table 3) with response options on a 5- point scale (1 = strongly disagree, 2 = disagree, 3 = neither disagree or agree, 4 = agree 5 = strongly agree). The SUS is a tool designed for assessing the usability of a product and has been normed across numerous platforms (e.g., Web sites, cell phones, TV applications). Scores range from 0 to 100. (SUS; Bangor, Kortum, & Miller, 2009)

CONTACTS AND LOCATIONS:
Overall Officials: Susan W Schroeder, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States